CLINICAL TRIAL: NCT05363267
Title: Study of Nutraceutical Intervention With High Phenolic Extra Virgin Olive Oil and Curcumin for Neurofibromatosis, Type 1 (NF1)
Brief Title: NF-1, Nutraceutical Intervention
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021LS032
Record Dates: First submitted 2022-04-26; First posted 2022-05-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Curcumin with high phenolic extra virgin olive oil (HP-EVOO) (Experimental): Identical for all participants with the exception of the curcumin dose level, which is assigned at study enrollment.
  Interventions: Dietary Supplement: curcumin, high phenolic extra virgin olive oil (HP-EVOO)

INTERVENTIONS:
Dietary Supplement: curcumin, high phenolic extra virgin olive oil (HP-EVOO) — identical for all participants with the exception of the curcumin dose level
  Dose 1: 1000 mg Curcumin daily dose with 1 capsule and 25 ml HP-EVOO volume at morning and night Dose 2: 2000 mg Curcumin daily dose with 2 capsules and 25 ml HP-EVOO volume at morning and night Dose 3: 4000 mg Curcumin daily dose with 4 capsules and 25 ml HP-EVOO volume at morning and night
  Other Names: curcumin; high phenolic extra virgin olive oil (HP-EVOO)

SUMMARY:
The treatment plan is identical for all participants with the exception of the curcumin dose level that is assigned at study enrollment. Participants are instructed to take the curcumin and olive oil one after the other (order does not matter) twice a day on an empty stomach ideally 30 minutes before breakfast and dinner.

Curcumin and high phenolic extra virgin olive oil (HP-EVOO) may continue for up to 12 months in the absence of unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* NF1 diagnosis based on NIH Consensus Conference Criteria and/or genetic testing
* Measurable cutaneous neurofibromas (cNFs) with or without plexiform NF
* Aged 18 years or older at the time of written consent
* Voluntary signed written consent obtained before the performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* Concurrent treatment with selumetinib or other MAPK, MEK or mTOR inhibitors, other targeted therapies, chemotherapy or radiation
* Conditions requiring systemic immunosuppression
* Swallowing difficulties or strong gag reflex which may interfere with study compliance
* Any comorbidities that may affect study participation in the judgement of enrolling investigator
* Psychiatric illness, cognitive challenges, social situations, or other circumstances that would limit compliance with study requirements, per judgment of the enrolling investigator
* Treatment with high phenolic olive oil or curcumin within six months of study entry
* Known pregnancy or anticipated conception during the 1 year study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to establish the safety and preliminary activity of curcumin and oleocanthal-rich olive oil supplementation in adult NF-1 persons with cutaneous neurofibromas. | End of treatment (12 months)
  The safety of this supplementation will be measured by the incidence of unacceptable/dose limiting toxicity (DLT) as defined any new Grade 2 or greater toxicity (based on CTCAE v 5).

SECONDARY OUTCOMES:
Characterize the toxicities associated with the planned intervention | 4 weeks after 1st dose of curcumin
  Incidence of unacceptable/dose limiting toxicity defined as any new ≥Grade 2 toxicity (based on CTCAE v 5) that cannot be attributed to the disease under treatment or other reason.
To evaluate the effect of the intervention on BMI | End of Treatment (12 months)
  The BMI will be measures across dose level group 95% confidence intervals.
To evaluate the effect of the intervention on lipid panel | End of Treatment (12 months)
  The lipid panel will be measures across dose level group 95% confidence intervals.
To assess the effect of the intervention on quality of life | End of treatment (12 months)
  Focused on skin related morbidity and pain will be evaluated using the average and range of SkinDex scale (0-100)
To determine preliminary efficacy of the intervention | End of treatment (12 months)
  Measure the volumetric measurement of target plexiform neurofibroma (% difference from baseline will be reported)
To identify issues with compliance to the planned intervention | End of treatment (12 months)
  Incidence of study deviations

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Moertel, MD, Principal Investigator — Masonic Cancer Center, Univeristy of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States